CLINICAL TRIAL: NCT05127291
Title: The Effect of Dual-Task on Hand Functions in Individuals With Type 2 Diabetes Mellitus
Brief Title: Dual-Task Effects on Hand Functions in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Eda Ozge OKUR, Assistant Proffessor, Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: T2DM-Dualtask
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; dual-task; hand functions
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients with type 2 diabetes mellitus
  Interventions: Other: Dual-task
- Control Group (Other): People without type 2 diabetes and prediabetes
  Interventions: Other: Dual-task

INTERVENTIONS:
Other: Dual-task — In the study, both groups are going to evaluate with and without dual-task. The dual-task will be counting back down 3 by 3 from a three-digit number.

SUMMARY:
The aim of the study is to examine the effect of dual-task performance on hand functions in individuals with Type 2 Diabetes Mellitus. It is planned to reach at least 100 participants during the data collection phase of the study. Demographic information, plasma glucose levels, and HbA1C levels of the participants included in the study will be recorded. The upper extremity problems of the participants will be recorded. Minnesota Manual Dexterity Test will be used to evaluate upper extremity functions.

DETAILED DESCRIPTION:
This study is aimed to evaluate the effect of dual-task performance on hand functions in individuals with Type 2 Diabetes Mellitus. The study will conduct in the Internal Medicine Clinic of Kutahya Health Sciences University Evliya Celebi Training and Research Hospital. Approval for the study was granted by the Clinical Research Ethics Committee of Kutahya Health Sciences University and written informed consent forms will be obtained from all the participants. This study is planned to reach at least 50 participants with type 2 diabetes mellitus for the study group and 50 participants without diabetes for the control group. The participants will be questioned about their eligibility for the inclusion criteria. The demographic and descriptive data of the participants will be recorded. Minnesota Manual Dexterity Test will be used to evaluate upper extremity functions. The test will be performed with and without the dual-task. Counting backward from a random three-digit number 3 by 3 will be used for the dual-task. The effect of dual-task will calculate using the difference between the completion time of both tests for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with type 2 diabetes mellitus for at least 5 years for study group, having no diagnosed type 2 diabetes mellitus or prediabetes for control group,
* Being able to count down 3 by 3 from a three-digit number,
* Volunteer to take part in the study.

Exclusion Criteria:

* History of traumatic or inflammatory injury in the upper extremity,
* History of involving the upper extremity in the last year,
* Having rheumatological/inflammatory arthritis or deformity,
* Having a deformity caused by osteoarthritis in the upper extremity,
* Having a neurological problem affecting the upper extremity,
* Getting 23 points or less on the Mini-Mental Test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The Minnesota Dexterity Test | 30 minutes
  The test consists of two parts, "placing" and "turning". The patient is instructed to put disks to the holes and the test time uses as a score, in the placing test. In the turning test, the patient is instructed to turn the disks before putting the holes. The test time is recorded. The test will perform with and without dual-task and the dual-task effect will calculate.
Dual-task effect | 30 minutes
  Each patient is going to be instructed to perform The Minnesota Dexterity Test with and without dual-task. Firstly, patients are going to perform the two parts of the test without dual-task. Secondly, patients are going to perform two parts of the test while counting down 3 by 3 from a random three-digit number. The percentage of difference is going to calculate as the dual-task effect.

CONTACTS AND LOCATIONS:
Overall Officials: Eda O Okur, Doctorate, Principal Investigator — Kutahya Health Sciences University; Ismail Okur, Doctorate, Study Director — Kutahya Health Sciences University; Turkan Pasali Kilit, Doctorate, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No